CLINICAL TRIAL: NCT00599222
Title: A Prospective, Randomized, Controlled Study on Intravitreal Ranibizumab (Lucentis) Combined With Transpupillary Thermotherapy (TTT) for Neovascular Age-related Macular Degeneration (AMD)
Brief Title: The Ranibizumab Plus Transpupillary Thermotherapy for Neovascular Age-Related Macular Degeneration (AMD) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anders Kvanta (Other)
Responsible Party: Sponsor-Investigator, Anders Kvanta, Professor, St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUTA001
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: AMD; macular degeneration; anti-VEGF; laser treatment
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TTT (Active Comparator): TTT is given every three months
  Interventions: Biological: ranibizumab; Procedure: TTT
- Sham TTT (Sham Comparator): Sham TTT is given every three months
  Interventions: Biological: ranibizumab; Procedure: Sham TTT

INTERVENTIONS:
Biological: ranibizumab — 0.5 mg intravitreal injection
  Other Names: Lucentis
Procedure: TTT — Transpupillary thermotherapy (TTT)
  Arms: TTT
Procedure: Sham TTT — Sham Transpupillary thermotherapy (TTT)
  Arms: Sham TTT

SUMMARY:
Neovascular age-related macular degeneration (AMD) is the leading cause of severe vision loss in the Western world. Intravitreal ranibizumab has recently become the treatment of choice for neovascular (AMD). Limitations to ranibizumab however include the high cost for the drug and the need for frequent intravitreal re-injections. The investigators' hypothesis is that when ranibizumab is combined with transpupillary thermotherapy (TTT) the number of necessary retreatments with Lucentis will be significantly reduced as compared to ranibizumab alone.

DETAILED DESCRIPTION:
Neovascular age-related macular degeneration (AMD) is caused by an ingrowth of pathological vessels under the macula. Experimental studies have demonstrated that vascular endothelial growth factor (VEGF) is centrally involved in this process. For this reason, anti-VEGF drugs, in particular ranibizumab, as become the treatment of choice for neovascular AMD. Ranibizumab use is limited by its high cost. Also, ranibizumab requires repeated (sometimes up to monthly) intravitreal injections for many years. Strategies to reduce the burden of this treatment on the patient as well as on the health care system will be critical. Combination therapy is an attractive such possibility. Transpupillary thermotherapy (TTT) is a technique by which vascular occlusion can be induced by delivering radiation at near infrared intensity to the target tissue through the pupil. Several reports have indicated that TTT may be used to slow disease progression in patients with neovascular AMD. In this study we examine whether combined ranibizumab and TTT will reduce the number of ranibizumab injections compared with ranibizumab alone (sham TTT). The study will go on for 2 years with an interim report after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* patients with subfoveal neovascular AMD with either classic/predominantly classic or occult lesions
* visual acuity => 20/200

Exclusion Criteria:

* subretinal fibrosis or atrophy under the fovea
* patients previously treated for neovascular AMD in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-02; Primary Completion 2009-11 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that will need 5 injections (loading phase excluded) or less with ranibizumab | 1 year

SECONDARY OUTCOMES:
Proportion of patients losing less than 15 letters on the ETDRS visual acuity chart | 1 year
Proportion of patients gaining more than 15 letters on the ETDRS visual acuity chart | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, Principal Investigator — St Eriks Eye Hospital
Locations (1):
- St Eriks Eye Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Soderberg AC, Algvere PV, Hengstler JC, Soderberg P, Seregard S, Kvanta A. Combination therapy with low-dose transpupillary thermotherapy and intravitreal ranibizumab for neovascular age-related macular degeneration: a 24-month prospective randomised clinical study. Br J Ophthalmol. 2012 May;96(5):714-8. doi: 10.1136/bjophthalmol-2011-300721. Epub 2012 Jan 12. PMID 22241923
- See also: Hospital homepage — http://www.sankterik.se